CLINICAL TRIAL: NCT01683279
Title: Pediatric Leukemia Adoptive Therapy (PLAT)-01: A Phase 1 Feasibility and Safety Study of Cellular Immunotherapy for Relapsed Pediatric CD19+ Acute Lymphoblastic Leukemia Using Autologous T-cells Lentivirally Transduced To Express a CD19-Specific Chimeric Antigen Receptor
Brief Title: A Pediatric Trial of Genetically Modified Autologous T Cells Directed Against CD19 for Relapsed CD19+ Acute Lymphoblastic Leukemia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Colleen Annesley, Medical Director, Seattle Children's Therapeutics, Seattle Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLAT-01
Record Dates: First submitted 2012-09-07; First posted 2012-09-11 (Estimated); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: B Cell Leukemia
Keywords: pediatric; acute lymphoblastic leukemia; CD19; Chimeric Antigen Receptor
MeSH Terms: conditions — Leukemia, B-Cell; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CAR+ T cells (Experimental): Subjects will receive two days of cyclophosphamide for a total of 3g/m^2 followed several days later by a single dose of Autologous CD19 CAR+ EGFTt + T cells
  Interventions: Biological: Autologous CD19 CAR+ EGFTt + T cells

INTERVENTIONS:
Biological: Autologous CD19 CAR+ EGFTt + T cells — Autologous T cell modified to express a CD19 specific CAR and a truncated EGFRt tag

SUMMARY:
Patients with relapsed leukemia often develop resistance to chemotherapy. For this reason, we are attempting to use a patient's own T cells, which can be genetically modified to expresses a chimeric antigen receptor(CAR). The CAR enables the T cell to recognize and kill the leukemic cells though the recognition of CD19, a protein expressed on the surface of the majority of pediatric ALL. This is a phase I study designed to determine the maximum tolerated dose of the CAR+ T cells and define the toxicity of the treatment. As a secondary aim, we will be looking at the efficacy of the T cells on eradicating the patient's leukemic cells.

DETAILED DESCRIPTION:
Upon meeting the eligibility requirements and enrolling on study, subjects will undergo a blood draw to obtain the T cells for the generation of the CD19 CAR+ T cells. The T cells are isolated from the blood, transduced with a lentivirus to express the CD19 CAR, and expanded in culture over a three week period. During the process of cell generation, subjects will continue to be cared for by their primary oncologist and may undergo additional treatment directed at the leukemia during this time.

After the CAR+ T cells have been generated, the subject undergoes a disease assessment and will be admitted to the hospital to receive 2 days of cyclophosphamide for lymphodepletion and reduction of disease burden. Several days later, the subject will receive an infusion of the CAR+ T cells.

Following treatment with the CAR+ T cells, subjects will be intensely followed for 6 weeks with serial blood testing and re-evaluation of disease status with bone marrow aspirates. After 6 weeks, the subjects clinical care will be resumed by their primary oncologist, and it is possible that they would receive additionally chemotherapy or a stem cell transplant.

Upon completion of the study, subjects will be followed at least annually with a either a medical history, physical exam and blood tests or a phone call/questionnaire for 15 years. This follow up will help to determine if the subject develops any long-term health problems related to the CAR+ T cells including a new cancer.

ELIGIBILITY:
Inclusion Criteria:

* CD19+ Leukemia in 1st marrow relapse with MRD at the end of 1st month of re-induction
* CD19+ Leukemia in 2nd or greater relapse
* CD19+ Leukemia with indication for HCT, but has contraindication
* Age between 1 and 26 years of age
* Karnofsky of >50 or Lansky >50
* Life Expectancy >12 weeks
* Able to tolerate a blood draw of 4-6mL/kg
* Recovered from acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy
* absolute lymphocyte count of >/=750 cell/mm3 or >/=500 is >20kg
* creatinine clearance or radioisotope GFR >/= 70mL/min/1.73m2 OR normal serum creatinine based on age/gender
* total bilirubin </= 1.5x upper limit normal OR direct bilirubin </= 1.5mg/dl
* ALT </= 3x upper limit normal
* corrected QTc <450msec of ECG
* Shortening Fraction >28% by ECHO or Ejection Fraction >50% by MUGA
* Documented negative HIV, Hep B and Hep C
* Agree to long-term follow up for up to 15 years if they receive T cell infusion

Exclusion Criteria:

* Philadelphia Positive Leukemia
* Prior Allogeneic Stem Cell Transplant
* CNS 2 or 3
* prior cellular immunotherapy with chimeric antigen receptor modified T cells
* fully humanized antibodies within three half lives
* systemic corticosteroids within 7 days of enrollment
* requires supplemental oxygen or has a chest X-ray with an infectious process
* CNS pathology (seizure disorder, paresis, aphasia, cerebrovascular ischemia/hemorrhage, severe brain injuries, dementia, cerebellar disease, organic brain syndrome, psychosis, coordination or movement disorder)
* Pregnant or breastfeeding women. Female participant of reproductive age must have a negative pregnancy test and agree to contraception for 1 year after T cell infusion.
* Active Malignancy other than CD19+ Leukemia
* Active severe infection defined as a positive blood culture within 48 hours of study enrollment or a fever >38.2C AND clinical signs of infection within 48 hours of study enrollment
* Patient has a concurrent medical condition, that in the opinion of the protocol PI or designee, would prevent the patient from undergoing protocol-based therapy.
* Trisomy 21
* Primary immunodeficiency/bone marrow failure syndrome

Ages: 1 Year to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2012-03-25 (Actual); Primary Completion 2015-01-07 (Actual); Study Completion 2030-01-07 (Estimated)

PRIMARY OUTCOMES:
Number of Participant with Adverse Events | 42 days
  The safety of the T cell infusion will be described and the maximum tolerated dose determined.

SECONDARY OUTCOMES:
Persistence of the CD19 CAR+ T cells | 42 days
  Patients will be followed for 42 days to determine if the transferred T cells remain detectable in the blood and bone marrow
Determine if there is anti-leukemic activity of the CD19 CAR+ T cells | 42 days
  Patients will have their bone marrow assessed following the T cell infusion to determine if their disease responded to the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Annesley, MD, Study Chair — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States